CLINICAL TRIAL: NCT01823692
Title: Study of Accuracy of Ultrasonography in Determining the Adequacy of Distal Radius Fracture Reduction
Brief Title: Evaluating Validity of Ultrasonography in Determining Distal Radius Fracture Reduction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Hamidreza Shemshaki, MD, Research Assistant, Isfahan University of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: ASD-1213-75
Record Dates: First submitted 2013-03-30; First posted 2013-04-04 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-03

CONDITIONS: Distal Radius Fracture
Keywords: Radius Fracture; Sensitivity; Reduction; Adequacy
MeSH Terms: conditions — Wrist Fractures; Radius Fractures; Hypersensitivity | interventions — High-Energy Shock Waves

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Distal Radius Fracture (Other): after manipulation and reduction were performed by single emergency medicine specialist under Bier block regional anesthesia or procedural sedation-analgesia, The ultrasonography was performed by the single emergency department physician in a long axis both in a anterioposterior and lateral views in determining whether the distal and proximal distal to a fracture was in a straight line (less than 3 mm difference) or not?
  Interventions: Other: ultrasonography

INTERVENTIONS:
Other: ultrasonography — after manipulation and reduction were performed by single emergency medicine specialist under Bier block regional anesthesia or procedural sedation-analgesia, The ultrasonography was performed by the single emergency department physician in a long axis both in a anterioposterior and lateral views in determining whether the distal and proximal distal to a fracture was in a straight line (less than 3 mm difference) or not?

SUMMARY:
The purpose of this study is to evaluate whether ultrasonography guidance compare with the simple radiography aids in determining the adequacy of distal radius fracture reduction.

DETAILED DESCRIPTION:
Distal radius fracture is one of the most common causes for visiting the emergency department. Nowadays, simple radiography is used as a control standard for evaluating reduction of distal radius fractures. The disadvantages include time wasting, frequent x-ray exposures and use of more sedation in determining adequate reduction, made scientists to evaluate alternative method such as ultrasonography which fast, easy and less dangerous were considered as advantages. The investigators goal was to identify whether ultrasonography guidance compare with the simple radiography aids in determining the adequacy of distal radius fracture reduction.

ELIGIBILITY:
Inclusion Criteria:

* > 21 years old and a diagnosing of a distal radius fracture based on simple radiography.

Exclusion Criteria:

* Open fractures
* more than 20 degree angulation
* joint internal involvement, communicated and along with Neurovascular compromised fractures
* patient's surgery due to other causes
* need to stay in the ICU and not being able to be treated at the same time for distal radius fracture
* patient's refusal to participate in the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2011-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
adequacy of distal radius fracture reduction | at 5 min after admission time
  after manipulation and reduction were performed by single emergency medicine specialist under Bier block regional anesthesia or procedural sedation-analgesia, The ultrasonography was performed by the single emergency department physician in a long axis both in a anterioposterior and lateral views in determining whether the distal and proximal distal to a fracture was in a straight line (less than 3 mm difference) or not?

CONTACTS AND LOCATIONS:
Overall Officials: Hamidreza Shemshaki, MD, Principal Investigator — Isfahan University of Medical Sciences
Locations (1):
- Al-Zahra University Hospital, Isfahan, Isfahan, Iran